CLINICAL TRIAL: NCT02565225
Title: Mobile Medically Supervised Patient Management in Rheumatoid Arthritis Patients Using DocuMed.rh and RheumaLive App
Brief Title: Mobile Medically Supervised Patient Management in Rheumatoid Arthritis
Acronym: MiDEAR
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: MiDEAR
Record Dates: First submitted 2015-09-16; First posted 2015-10-01 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- RheumaLive App use: RheumaLive App use and evaluation of feasibility
  Interventions: Behavioral: RheumaLive App use
- RheumaLive App use & threshold values: RheumaLive App use and evaluation of feasibility
  Interventions: Behavioral: RheumaLive App use

INTERVENTIONS:
Behavioral: RheumaLive App use

SUMMARY:
The purpose of this study is to evaluate the use, usability and feasibility of an Application (App) for patients with rheumatoid arthritis with diary functionalities, in patient-physician interaction.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years, owner of App capable device, RA, informed consent

Exclusion Criteria:

* non German speaking, no App capable device available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of use of the RheumaLive Application in patients with rheumatoid arthritis. | baseline and change over up to nine months
  Evaluation of use by counting and by a patient paper-based questionnaire

SECONDARY OUTCOMES:
Comparison paper-based vs electronic PROM in the App - Differences of the scores | baseline and change after 3 months
  RADAI - Rheumatoid Arthritis Disease Activity Index and FFbH (Hannover Functional Ability Questionnaire ) / calculated HAQ (Health Assesment Questionnaire)
Evaluation of feasibility of the RheumaLive Application in patients with rheumatoid arthritis. | at 3 months from start and change over 6 more months
  Evaluation of feasibility by a patient and a physician paper-based questionnaire
Evaluation of usability of the RheumaLive Application in patients with rheumatoid arthritis. | at 3 months from start and change over 6 more months
  Evaluation of usability by a patient paper-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schneider, Prof., Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (1):
- Policlinic for Rheumatology & Hiller Research Centre for Rheumatology, Düsseldorf, Germany

REFERENCES:
- [Derived] Richter JG, Nannen C, Chehab G, Acar H, Becker A, Willers R, Huscher D, Schneider M. Mobile App-based documentation of patient-reported outcomes - 3-months results from a proof-of-concept study on modern rheumatology patient management. Arthritis Res Ther. 2021 Apr 19;23(1):121. doi: 10.1186/s13075-021-02500-3. PMID 33874994